CLINICAL TRIAL: NCT04568135
Title: A Survey Study to Assess the Impact of the COVID-19 Pandemic on Participants With Pre-Existing Mental Health Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Siyan Clinical Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: SCR-SUR-001
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: survey; covid19; Pre-Existing Mental Health Diagnosis
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- survey
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — survey

SUMMARY:
The primary objective of this survey study is to assess the impact of the current COVID-19 pandemic on participants with psychiatric disorders to identify areas of needed support and services. Data collected may serve as a foundational research in the prevention, care and treatment of mental health disorders during pandemics such as COVID-19. This survey study will utilize the Epidemic-Pandemic Impacts Inventory (EPII). This is a newly tool designed to assess tangible impacts of epidemics and pandemics across personal and social life domains.

DETAILED DESCRIPTION:
This study is a survey study designed to assess the impact of the current COVID-19 pandemic on participants with psychiatric disorders to identify areas of needed support and services. This survey is an exploratory investigation of patient experience to guide Siyan in program improvement and development of next steps to serve patients. A one-time survey will be sent out electronically via email to approximately 3,500 adult patients in the Siyan Clinical Corporation and Siyan Clinical Research practices. The survey will consist of the Epidemic-Pandemic Impacts Inventory (EPII). This is a new tool designed to assess tangible impacts of epidemics and pandemics across personal and social life domains.

Siyan staff will derive a list of patients from the Siyan EHR who meet eligibility criteria. The list will include Patient ID, age, gender, ethnicity, occupation, employment status, primary diagnosis, and last known email address. Each patient in the sample will receive an email inviting them to participate in the survey, explaining the purpose of the survey, how Siyan will use the survey results, and how the survey will be administered. All patients in the sample who have not responded will also receive a reminder email approximately one week later. Each e-mail will include information to contact the Investigator with any questions.

Patients that reply to the initial invitation will receive the electronic Informed Consent Form (eICF) to sign and return to the Project Coordinator via Adobe Sign. The Project Coordinator will track the name and email address of all patients who consent to participate, and will send each a link to the online survey in SurveyGizmo. https://www.surveygizmo.com/s3/5751791/Siyan-COVIDImpactSurvey) The online survey will repeat the text of the electronic Informed Consent Form (eICF), allowing participants to again confirm agreement and continue the survey or disagree and exit out. Participants who agree to the consent will be asked to confirm their email address, and respond to the 92 questions in the EPII about how the coronavirus disease pandemic has changed their and/or their family's lives. Respondents will also be asked basic demographic questions: age, gender identity, ethnicity, education level, employment status, industry, children under 18 in the home, marital status, and experience with basic psychiatric disorders.

The evaluation consultant will tabulate responses and provide basic frequencies and analyses to the Investigator, along with a de-identified dataset for further advanced analysis. Data collected may serve as a foundational research in the prevention, care and treatment of mental health disorders during pandemics such as COVID-19. Analysis of data collected will be published in academic journals to serve as a foundational research in the prevention, care and treatment of mental health disorders during pandemics such as COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agrees to participate in the study under their own free will and is willing/able to agree to an informed e-consent form indicating that he/she understands the purpose of the study, the procedures that are required for the study, and that he/she is willing to participate in the study.
* Female or male and between the ages of 18 and 80, inclusive at the time of consent.
* Is a currently receiving or has previously received psychiatric services from Siyan Clinical Corporation and/or Siyan Clinical Research practices.
* Is capable of understanding and complying with study requirements.
* Has agreed to the e-ICF. No study-related procedures will be performed before the participant has agreed to the consent letter.

Exclusion Criteria:

* A known diagnosis of dementia will not be included in the sample.
* Under the age of 18 or over the age of 80.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a survey study designed to assess the impact of the current COVID-19 pandemic on participants with psychiatric disorders to identify areas of needed support and services. This survey is an exploratory investigation of patient experience to guide Siyan in program improvement and development of next steps to serve patients.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Survey: Epidemic-Pandemic Impacts Inventory (EPII) | one year
  The Epidemic-Pandemic Impacts Inventory (EPII) is a newly tool designed to assess tangible impacts of epidemics and pandemics across personal and social life domains. Candidate items were constructed by a team of clinical and developmental psychologists with expertise in assessment of stress, trauma, resilience, and coping. Feedback from professionals across multiple disciplines (e.g., social work, pediatrics, medicine, anthropology) was incorporated in selecting and refining final items for of the measure, which was accomplished via expert consensus.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah A, Darling M, Arstein-Kerslake O, Morgan T, Vance Tovrea A, Young J, Laines H. Measuring the Impact of COVID-19 on Siyan Mental Health Patients Using the Epidemic-Pandemic Impacts Inventory: Survey Study. JMIR Form Res. 2021 Jul 29;5(7):e29952. doi: 10.2196/29952. PMID 34323851